CLINICAL TRIAL: NCT01331278
Title: A Comparative Study of Knee Systems Employing Personalized Computer Generated Cutting Guides for Total Knee Arthroplasty
Brief Title: A Comparative Study of Knee Systems
Acronym: Bake-Off
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Foundation for Southwest Orthopedic Research (Other)
Responsible Party: David R. Lionberger, MD, Southwest Orthopedic Group, LLP
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0509-0060
Record Dates: First submitted 2011-04-06; First posted 2011-04-08 (Estimated); Last update posted 2011-04-08 (Estimated); Status verified 2011-04

CONDITIONS: Osteoarthritis of the Knee
Keywords: total joint replacement; knee
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Arthroplasty, Replacement, Knee

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Custom Cutting Blocks (Active Comparator)
  Interventions: Procedure: Total Knee Arthroplasty with Custom Cutting Blocks
- Computer Assisted Surgery (Active Comparator)
  Interventions: Procedure: Total Knee Arthroplasty via Computer Assisted Surgery

INTERVENTIONS:
Procedure: Total Knee Arthroplasty with Custom Cutting Blocks — Subjects randomized to this study group will undergo TKA with patient specific custom cutting blocks generated by pre-op MRI and a Biomet Vanguard knee implant
  Other Names: Signature Knee System
  Arms: Custom Cutting Blocks
Procedure: Total Knee Arthroplasty via Computer Assisted Surgery — Subjects randomized to this study group will receive TKA via computer assisted surgery and a Biomet Vanguard knee implant
  Arms: Computer Assisted Surgery

SUMMARY:
The custom cutting guides personalized for each patient via pre-operative MRI will result in significantly faster intraoperative time with comparable knee alignment accuracy, cost, knee function, and patient satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* must be scheduled to undergo TKA with no bilateral TKA planned within 6 weeks of the initial surgery date
* must be 18 years of age or older
* must be capable and willing to provide informed consent
* must have flexion contracture less than 15 degrees.
* must have ligament stability no more than 2 degrees instability in varus/valgus extension stress

Exclusion Criteria:

* medical condition or personal circumstances that will prevent participation and completion of the follow-up visits at 3 weeks, 6 weeks and 3 months post-op
* currently participating in or has participated in (within 30 days prior to inclusion in this study) another clinical trial of an investigational drug, biologic, device, or procedure
* known pre-operative systemic infections, uncontrolled diabetes, or diseases or conditions that are known to interfere with the wound healing process
* Knee alignment deformities greater than 7 degrees varus or valgus
* known prior knee revisions or previous surgeries deemed to compromise the TKA incision exposure
* known medical conditions prohibiting the use of MRI or nickel allergy, sensitivity, or hardware in the region of the knee

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2009-09; Primary Completion 2010-08 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
mean intraoperative time | measured during surgery (day 1)
  Time measured in pre-defined segments from the point that the patient is wheeled into the OR until the OR is clean and ready for the next case's activities to begin.

SECONDARY OUTCOMES:
alignment accuracy | 3 weeks post-op

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Southwest Orthopedic Group, LLP, Houston, Texas
  - The Methodist Hospital, Houston, Texas

REFERENCES:
- [Derived] Lionberger DR, Crocker CL, Chen V. Patient specific instrumentation. J Arthroplasty. 2014 Sep;29(9):1699-704. doi: 10.1016/j.arth.2014.03.019. Epub 2014 Mar 28. PMID 24810539